CLINICAL TRIAL: NCT02065505
Title: METHOD PILATES x PILATES IN WATER POSTURAL ALIGNMENT AND ITS CORRELATION WITH RESPIRATORY CAPACITY WITH HEMIPARESIS SPASTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19284013.6.0000.5503
Record Dates: First submitted 2014-02-07; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
Keywords: Spastic hemiparesis; Posture; Pilates; Respiratory Capacity
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilates Group Solo (Experimental): participate in this group 30 individuals who will be treated with the Pilates Method performing the exercises on the ground, using the Swiss ball and elastic bands. The exercises will aim to lengthen the musculature that are shortened due to the characteristic postural pattern of pathology (major and minor pectoral, shoulder adductors, biceps, wrist flexors, trunk side chain); strengthen the musculature that provide postural support (abdominal, middle trapezius, rhomboids, gluteus maximus, erector spinae and latissimus dorsi) and the upper limb musculature important for activities of daily living (triceps, biceps, internal rotators, external rotators and abductors of the shoulder).
  Interventions: Other: Mat Pilates
- Water Pilates Group (Experimental): participate in this group 30 individuals who will be treated with the Pilates method, but doing the exercises in the therapy pool, with the aid of floats and weights. The protocol of stretches and exercises will work the same muscle groups than the G1, keeping the same decubitus whenever possible. The adaptations to the exercises are justified by the physical principles of water, which at one point may act for or against the activity being performed.
  Interventions: Other: Water Pilates

INTERVENTIONS:
Other: Mat Pilates
  Arms: Pilates Group Solo
Other: Water Pilates
  Arms: Water Pilates Group

SUMMARY:
To evaluate the efficacy of treatment with the Pilates Method in postural alignment and its correlation with the respiratory capacity of individuals with hemiparesis, with the aid of biomedical instrumentation, comparing the method performed in soil and therapy pool.

DETAILED DESCRIPTION:
The hemiparesis, which corresponds to muscle weakness in hemisphere contralateral to injury, is the most common disorder after stroke Brain. The most obvious implication is postural asymmetry, having direct relation to respiratory pressures are also reduced due to muscle weakness, thus altering the respiratory capacity of these individuals. The Pilates Method is gaining prominence in clinical and scientific areas, contributing to restoring good posture and vertical alignment of the body. Therefore, this study aims assess muscle electrical activity, respiratory capacity and functionality of spastic hemiparetic patients before and after application the Pilates Method, soil and therapy pool. A randomized study where 60 hemiparetic participate will be held with brachial predominance and 30 healthy subjects (Control Group), of both sexes, ages 40 to 70 years. Individuals with hemiparesis will be randomly assigned through a lottery and half held 10 consecutive sessions of Pilates in the soil and the rest will the same protocol adapted for therapy pool. The control group will be treated by the Pilates Method in the soil. The exercises will aim to lengthen musculature shortened due to postural pattern of pathology ; strengthen selected muscles that give support and postural musculature more important upper limb for activities of daily living. Participants will undergo postural assessment, activity EMG, muscle strength, respiratory capacity analysis and evaluation of the functionality of the upper limbs on the first day of treatment and after doing all sessions. The Student's t test will be used, with a significance level of 5 % to compare results obtained before and after treatment. After the tests, the Pearson correlation will also be made between the data obtained in soil and therapy pool. Thus, it is expected that Pilates can improve postural alignment and the breathable hemiparetic and the strengthening of specific muscles of the upper limbs assist in improving the functionality of them in their daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered cerebrovascular accident for at least two years (chronic hemiparesis) with prevalence of upper limb (middle cerebral artery);
* Spasticity grade 1, 1 + 2 by the Modified Ashworth Scale;
* Good cognition;
* Get assume a standing position
* Sign the Consent form;

Inclusion Criteria for Healthy individuals who will make up the control group:

* People who may be standing upright;
* Understand the activities that will be proposed
* Subscribe to the disclaimer conscentimento.

Exclusion Criteria:

* Patients with severe cardiovascular disease;
* Patients with joint deformities;
* Patients with balance disorders;
* Patients with seizures;
* Patients with hypertension;
* Patients with uncontrolled diabetes;
* Individuals with a restriction in the liquid medium;
* Individuals with cognitive impairment that prevents an understanding of the proposed activities.

Exclusion criteria for the control group:

* Individuals who do not meet the age range studied;
* Patients with uncontrolled hypertension and diabetes;
* Individuals with restrictions on liquid medium;
* Subjects with any neurological disorder;
* Individuals with severe respiratory diseases;
* Individuals who have been diagnosed with severe postural imbalance.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
muscle electrical activity before and after treatment | 4 weeks
  The electrical activity of the postural muscles will be measured before and after treatment.

SECONDARY OUTCOMES:
respiratory capacity before and after treatment | 4 weeks
  Will be measured respiratory capacity of the participants (tidal volume, residual volume, etc.) before and after treatment.
higher functionality members before and after treatment | 4 weeks
  Will be measured through a range of functionality, the functionality of the upper limbs of the subjects, seeking an improvement in their activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Engineering Laboratory of Sensory Motor, São José dos Campos, São Paulo, Brazil